CLINICAL TRIAL: NCT03126162
Title: A Randomized, Controlled Trial Evaluating 2 Techniques of Postoperative Bladder Testing for Patients Undergoing Same-day Total Laparoscopic Hysterectomy
Brief Title: Postoperative Bladder Testing After Total Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Suketu Mansuria, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PRO17010292
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Laparoscopic Hysterectomy; Enhanced Recovery After Surgery
Keywords: minimally invasive gynecologic surgery; same-day discharge; bladder testing

STUDY DESIGN:
Intervention Model Description: A randomized, controlled trial evaluating 2 techniques of postoperative bladder testing for patients undergoing same-day total laparoscopic hysterectomy
Who Masked: Participant
Masking Description: Participants will be randomly assigned to one of two groups - A) bladder backfilled group or B) control group. This is a blinded study and the participant will not know which group they were assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bladder Backfilled group (Experimental): Subjects randomized to the bladder backfilled group (Group A) will have 200 mL of normal saline instilled into their bladders prior to removal of the foley catheter. The foley catheter will subsequently be removed
  Interventions: Procedure: InstilIing normal saline into bladder; Procedure: Removal of foley catheter
- Control group (Placebo Comparator): Subjects randomized to the control group (Group B) will just have their foley catheters removed at the end of the surgery. This is routinely done post-operatively after routine gynecologic surgery.
  Interventions: Procedure: Removal of foley catheter

INTERVENTIONS:
Procedure: InstilIing normal saline into bladder — Backfilling the bladder with 200 mL of normal saline immediately postoperatively, prior to foley catheter removal, after same-day total laparoscopic hysterectomy can potentially increase time to first spontaneous void and time to discharge.
  Arms: Bladder Backfilled group
Procedure: Removal of foley catheter — Removal of the foley catheter is routinely performed after same-day laparoscopic hysterectomy

SUMMARY:
The objective of this study is to determine if backfilling the bladder immediately post-operatively, prior to removal of the foley catheter, in patients undergoing same-day total laparoscopic hysterectomy will hasten time to first spontaneous void and time to discharge

DETAILED DESCRIPTION:
In recent years, a paradigm shift from traditional perioperative care models to "Enhanced Recovery After Surgery (ERAS)" has taken place across a wide range of surgical subspecialties including minimally-invasive gynecologic surgery. Many gynecologic procedures that once required hospital admission are now being performed as outpatient procedures. To optimize same-day discharge through the ERAS pathways, protocols call for early removal of urinary catheters following gynecologic surgery. Studies in urogynecologic literature have shown that a backfill-assisted voiding trial is superior to a spontaneous voiding trial in patients undergoing transvaginal surgery. However, there are limited studies published in literature focusing on minimally invasive gynecologic procedures, specifically laparoscopic hysterectomies. A successful spontaneous voiding trial is usually a postoperative criteria prior to discharge after same-day total laparoscopic hysterectomy. Through this randomized controlled trial, the investigators aim to compare two techniques of postoperative bladder testing for patients undergoing same-day total laparoscopic hysterectomy. This study would provide valuable data on improved measures for predicting voiding efficiency, time to first void, and time to discharge for patients undergoing same-day total laparoscopic hysterectomies. Ultimately, the investigators predict that backfilling the bladder immediately postoperatively, prior to removal of the foley catheter, will hasten time to first spontaneous void and reduce the amount of time spent in the recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-75 years of age
* Ability to comprehend English
* Women undergoing same-day laparoscopic hysterectomy through the Enhanced Recovery after Surgery (ERAS) protocol at Magee-Womens Hospital (includes total laparoscopic hysterectomy, laparoscopic supracervical hysterectomy, laparoscopic-assisted vaginal hysterectomy)

Exclusion Criteria:

* Women who are unable to give informed consent
* History of prior or concurrent urogynecologic procedures performed including mid-urethral sling, rectocele/cystocele repairs, burch urethropexy, sacrospinous ligament fixation, uterosacral vaginal vault suspension, sacrocolpopexy
* History of multiple sclerosis
* Known malignancy of the bladder
* Bladder or ureteral injury that occurred intra-operatively
* Women who are being treated for an active urinary tract infection at the time of surgery
* Women admitted overnight who fail to go home the same day after total laparoscopic hysterectomy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Hysterectomies are only performed on women.
Enrollment: 172 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2018-05-04 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Time to first spontaneous void | From the date of randomization until the date of discharge from the hospital, assessed up to 4 weeks
  Our primary hypothesis is that patients who undergo same-day total laparoscopic hysterectomy that are randomized into the group who have their bladders backfilled with 200 cc normal saline post-operatively, prior to removal of the foley catheter will have a shorter time to first spontaneous void.

SECONDARY OUTCOMES:
Time to discharge from the hospital after same-day laparoscopic hysterectomy | From the date of randomization until the date of discharge from the hospital, assessed up to 4 weeks
  We hypothesize that patients who undergo same-day total laparoscopic hysterectomy that are randomized into the group who have their bladders filled with 200 cc normal saline post-operatively, prior to removal of the foley catheter, will have a shorter time to discharge. We will be recording the amount of time patients spend in the post-anesthesia care unit (PACU)

OTHER OUTCOMES:
Post-operative urinary retention rates | From the date of randomization until the date of discharge from the hospital, assessed up to 4 weeks
  We will also evaluate the rates of postoperative urinary retention in patients who undergo same-day total laparoscopic hysterectomy through the Enhanced Recovery After Surgery (ERAS) protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Suketu Mansuria, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Magee-Womens Hospital, UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Authorized representatives of Magee-Womens Hospital of UPMC may have access to research data/documents for the purpose of research. These 'external persons' may include other investigators from both inside and outside Magee-Womens Hospital of UPMC who are conducting similar research after IRB approval. The data that would be shared would be de-identified research data/materials. The investigators currently do not have a data sharing plan with individuals other than the current investigators/research staff involved with this research project. Should the investigators decide to share data in the future, the investigators will contact the Office of Research before sharing de-identified research data/materials to determine whether an agreement needs to be executed.

REFERENCES:
- [Result] Kalogera E, Dowdy SC. Enhanced Recovery Pathway in Gynecologic Surgery: Improving Outcomes Through Evidence-Based Medicine. Obstet Gynecol Clin North Am. 2016 Sep;43(3):551-73. doi: 10.1016/j.ogc.2016.04.006. PMID 27521884
- [Result] Modesitt SC, Sarosiek BM, Trowbridge ER, Redick DL, Shah PM, Thiele RH, Tiouririne M, Hedrick TL. Enhanced Recovery Implementation in Major Gynecologic Surgeries: Effect of Care Standardization. Obstet Gynecol. 2016 Sep;128(3):457-66. doi: 10.1097/AOG.0000000000001555. PMID 27500337
- [Result] Kalogera E, Bakkum-Gamez JN, Jankowski CJ, Trabuco E, Lovely JK, Dhanorker S, Grubbs PL, Weaver AL, Haas LR, Borah BJ, Bursiek AA, Walsh MT, Cliby WA, Dowdy SC. Enhanced recovery in gynecologic surgery. Obstet Gynecol. 2013 Aug;122(2 Pt 1):319-328. doi: 10.1097/AOG.0b013e31829aa780. PMID 23969801
- [Result] Foster RT Sr, Borawski KM, South MM, Weidner AC, Webster GD, Amundsen CL. A randomized, controlled trial evaluating 2 techniques of postoperative bladder testing after transvaginal surgery. Am J Obstet Gynecol. 2007 Dec;197(6):627.e1-4. doi: 10.1016/j.ajog.2007.08.017. PMID 18060956
- [Derived] Chao L, Mansuria S. Postoperative Bladder Filling After Outpatient Laparoscopic Hysterectomy and Time to Discharge: A Randomized Controlled Trial. Obstet Gynecol. 2019 May;133(5):879-887. doi: 10.1097/AOG.0000000000003191. PMID 30969209